CLINICAL TRIAL: NCT07161466
Title: The Influence of Different PEEP Levels After Recruitment Maneuvre on the Effect of Alveolar Recruitment Maintenance and Patients' Cardiac Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Study Director, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024ky380
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: PEEP=0 cmH2O (Experimental): After the patient enters the operating room, routine monitoring of ECG, non-invasive blood pressure, and SpO₂ is performed. Followed by radial artery cannulation for invasive arterial blood pressure monitoring.Then connect the Weijie FloTrac Cardiac Output Monitoring Device.
  After 3 minutes of pre-oxygenation, tracheal intubation is performed with the following ventilation parameters: VT 6-8 ml/kg, FiO₂ 60%, RR 15 breaths/min, I/E 1:2, and PEEP 4 cmH₂O. Ten minutes after the establishment of pneumoperitoneum during the surgery, baseline levels of respiratory mechanics parameters and hemodynamic variables are recorded. Subsequently, alveolar recruitment is performed at a pressure of 30 cmH₂O for 30 seconds. Immediately after recruitment, the PEEP level is adjusted to 0 cmH2O. The changes in respiratory mechanics parameters and hemodynamic variables after recruitment are recorded. After the outcome indicators recover to the new baseline level, the PEEP is readjusted to 4 cmH₂O.
  Interventions: Behavioral: lung recruitment maneuvre; PEEP
- B: PEEP=4cmH2O (Experimental)
  Interventions: Behavioral: lung recruitment maneuvre; PEEP
- C: PEEP=8cmH2O (Experimental)
  Interventions: Behavioral: lung recruitment maneuvre; PEEP
- D: PEEP=12cmH2O (Experimental)
  Interventions: Behavioral: lung recruitment maneuvre; PEEP

INTERVENTIONS:
Behavioral: lung recruitment maneuvre; PEEP — After the patient enters the operating room, routine monitoring of ECG, non-invasive blood pressure, and SpO₂ is performed. Local anesthesia is used for radial artery puncture and catheterization to monitor invasive blood pressure.
  After 3 minutes of pre-oxygenation, tracheal intubation is performed with the following ventilation parameters: VT 6-8 ml/kg, FiO₂ 60%, RR 15 breaths/min, I/E 1:2, and PEEP 4 cmH₂O. Ten minutes after the establishment of pneumoperitoneum during surgery, baseline levels of respiratory mechanical parameters and hemodynamic variables are recorded. Subsequently, alveolar recruitment is performed at a pressure of 30 cmH₂O for 30 seconds. Immediately after recruitment, the PEEP level is adjusted according to the group. The changes in respiratory mechanics parameters and hemodynamic variables after recruitment are recorded. After the outcome indicators recover to the new baseline level, the PEEP is readjusted to 4 cmH₂O.

SUMMARY:
During general anesthesia surgery, the role of positive end-expiratory pressure (PEEP) in mechanical ventilation remains uncertain. Pressure levels above 0 cm H₂O can prevent postoperative pulmonary complications but may also cause intraoperative circulatory depression and lung injury due to overdistension. Using very low levels of PEEP may lead to atelectasis. However, high levels of PEEP can not only trigger complications such as intraoperative circulatory depression but also promote hyperinflation. Positive end-expiratory pressure (PEEP) is required to prevent atelectasis during lung-protective ventilation, and different levels of PEEP exhibit varying physiological and clinical effects when used alone or in combination with alveolar recruitment maneuvers (ARM). Alveolar recruitment maneuvers (ARM) are used to open atelectatic lung parenchyma, but the duration of their benefits has not been clearly determined. This study aims to determine the effectiveness of different PEEP levels after ARM in general anesthesia surgery, the duration of their time-dependent responses, and their hemodynamic effects, providing a reference for how often recruitment maneuvers should be performed during general anesthesia and further refining the specific details of lung-protective ventilation strategies.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classification: Ⅰ or Ⅱ or Ⅲ
* Adults aged 18 to 80 years, regardless of gender.
* Patients undergoing elective laparoscopic surgery under general anesthesia.
* Patients who have provided written informed consent after understanding the study purpose, procedures, and potential risks.

Exclusion Criteria:

* Recent thoracic surgery; chest X - ray or CT indicating pneumothorax, emphysema, or pulmonary bullae;
* Pulmonary diseases: asthma, severe obstructive ventilatory dysfunction; preoperative pulse oxygen saturation (SpO2) < 90% in room air or SpO2 < 95% with oxygen supplementation; contraindications for lung recruitment: high intracranial pressure, hypovolemic shock, right heart failure;
* Severe heart disease (New York Heart Association, NYHA Class III or IV; acute coronary syndrome or sustained ventricular tachyarrhythmia); participation in other interventional studies or refusal to be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
the duration of improvement in lung compliance | during the surgery

IPD SHARING:
Plan to Share IPD: No